CLINICAL TRIAL: NCT05963399
Title: An Integrated Care Platform Based on the Monitoring of Older Individual Intrinsic Capacity for Inclusive Health (CAREUP)
Acronym: CAREUP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INRCA_007_2023
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Old Age
Keywords: ageing; older adults; artificial intelligence; informal caregiver; usability; acceptance; Intrinsic capacity; quality of life; wellbeing; loneliness; ICT-based solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- older adults (Experimental): Elderly adults who live independently in their own home in rural or urban areas.
  Interventions: Device: CAREUP platform

INTERVENTIONS:
Device: CAREUP platform — The Experimental Group will test the CAREUP platform at home for 12 months.

SUMMARY:
The objective of this study is to assess the usability and acceptance of the CAREUP solution in improving the quality of life at home of the older adults. The CAREUP solution is a platform that collects data from different tools such as tablets, smartwatches, ambient sensors, iHealth weight scale, and Digital Hand Dynamometer.

.

DETAILED DESCRIPTION:
The objective of this study is to assess the usability and acceptance of the CAREUP solution at home in primary (older adults), secondary (informal caregivers) and tertiary (doctors and geriatrics) end users. The CAREUP solution is a platform that collects data from different tools such as tablets, smartwatches, ambient sensors, iHealth weight scale, and Digital Hand Dynamometer. The study will comprehends two phases: a pre-pilot and pilot phases.The pre-pilot phase will test new user interfaces and games with 5 older adult (primary users) and 5 informal caregiver (secondary) in each site (Italy, Romania, Austria) for at least 1 week. This phase will only focus on primary endpoints (usability and acceptance). The pilot phase will investigate platform usability, acceptance and efficiency of developed Intrinsic Capacity (IC) evaluation algorithms, reliability and security. At least 30 primary and 15 secondary and some tertiary users (doctors and geriatrics) will be enrolled in each country (Italy, Romania, Austria) for 12 months. This phase will focus on both primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Live independently in their home in rural or urban areas;
* In good physical and cognitive status;
* Able to stand and walk unaided;
* Availability to sign the Informed Consent;
* Ability to use smartphones/tablets independently.

Exclusion Criteria:

* Use of active implant or not-implant medical devices;
* Allergy to nickel components;
* Lack of written informed consent;
* Acute or untreated medical problems such as history of syncopal episodes, epilepsy and vertigo not controlled pharmacologically; serious dysfunction of the autonomic system; severe behavioural syndromes not compensated by drugs; concurrent neurological diseases; severe systemic diseases with life expectancy < 1 year;
* A myocardial infarction or stroke within 6 months;
* Painful arthritis, spinal stenosis, amputation, painful foot lesions or neuropathy limiting balance and mobility;
* Uncontrolled hypertension;
* Pacemaker or implantable cardioverter defibrillator;
* Diagnosis of mild and or/advanced Parkinson's disease or other neuromuscular disorder;
* Diagnosis of mild and/or advance cognitive impairments
* Metastatic cancer or immunosuppressive therapy;
* Significant visual or hearing impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-12-14 (Estimated); Study Completion 2024-12-14 (Estimated)

PRIMARY OUTCOMES:
Change in acceptability of the CAREUP platform | baseline and 12 months later
  Acceptability will be assess by an ad hoc structured questionnaire of 10 questions to collect data about like and dislike of the Careup platform.
Change in usability of the CAREUP platform | baseline and 12 months later
  The System Usability Scale (SUS) is a reliable tool for measuring usability. It consists of a10 item questionnaire with five response options for respondents from 'Strongly agree' to 'Strongly disagree'.

SECONDARY OUTCOMES:
Change in Physical Performance | baseline, 6 and 12 months later
  Short Physical Performance Battery (SPPB) is a short battery of tests designed to assess the function of the lower limbs. This scale consists of 3 different sections: balance assessment, evaluation of walking on 4 linear meters, evaluation of the ability to perform, for 5 consecutive times, the sit to stand from a chair, without using the upper limbs. The total scale score therefore has a range from 0 to 12. A total score below 10 indicates frailty and a high risk of disability and falls. The 1-point change in score from pre to post test is of clinical relevance.
Change in Quality of Life | baseline, 6 and 12 months later
  The EuroQol-5D-5L (EQ-5D-5L) scale consists of five dimensions: mobility, independence, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, mild problems, moderate problems, severe problems and extreme problems. The participant is asked to indicate his/her health status by ticking the box corresponding to the most appropriate statement in each of the five dimensions. The numbers from the five dimensions can be combined into a 5-digit number that describes the health status of the participant. The numerals 1-5 have no arithmetic properties and should not be used as a cardinal score. In addition, there is the EQ Visual Analogue scale (EQ VAS).The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. The EQ-5D-5L now asks respondents to simply 'mark an X on the scale to indicate how your health is TODAY'.
Change in Mood | baseline, 6 and 12 months later
  The 15-item Geriatric Depression Scale (GDS-15) assesses the current condition of the patient's mood. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Stara, Study Chair — IRCCS INRCA, Ancona, Italy
Locations (3):
- EURAG Austria, Vienna, Austria
- IRCCS INRCA Hospital, Ancona, Italy
- Ana Aslan International Foundation, Bucharest, Romania